CLINICAL TRIAL: NCT03006549
Title: Using Emergency Manuals During Interprofessional Crisis Management: Are There Unintended Consequences?
Acronym: EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Richard D Urman, Associate Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P000133
Record Dates: First submitted 2016-12-23; First posted 2016-12-30 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Safety Issues
Keywords: Emergency Manual; Crisis Checklist

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emergency Manual (Experimental): emergency manual present
  Interventions: Behavioral: Emergency Manual (Crisis Checklist)
- No Emergency (No Intervention): NO emergency manual present

INTERVENTIONS:
Behavioral: Emergency Manual (Crisis Checklist) — participants will have an Emergency Manual available to them during the crisis simulation scenario.
  Arms: Emergency Manual

SUMMARY:
Despite increasing interest in emergency manuals (EMs), relatively little is known about their effectiveness and limitations in the perioperative setting. Prior studies have been limited in that they evaluated EMs using crises that were tailor-made to match one of their chapters, and there has been minimal participation by attending surgeons and other experienced personnel. The Investigators' preliminary experience suggests less-than-expected EM use and suboptimal usage, which may be due to the simulation scenario falling "halfway between" two different chapters of the EM, raising the question of whether limitations were due to the EM content, team dynamics, or inadequate training in the EM use. In this randomized, prospective, two-center simulation-based study, the investigators utilize clinical scenarios specifically designed to observe the patterns of use and to test the limitations of the EMs. The hypothesis is that EMs may not improve, and may even worsen, clinical performance in situations that do not exactly match a specific chapter of that EM, and that EM usage patterns will identify both strengths and limitations of the tools and its implementation. The participating healthcare providers consisting of experienced surgeons, anesthesiologists, and nurses will be randomized into four experimental groups, each exposed to either a "specific" or "non-specific" simulation scenario, along with or without the availability of the EM. The major experimental endpoint will be how many "critical actions" each team performs, scored as the percentage of actions taken from a pre-determined list. The goal of this study is to improve EM content and use by understanding its limitations during interprofessional team-training simulations and to study whether EMs enhance or detract from clinical performance. This is especially a concern in situations that do not exactly match a specific chapter of the EM, such as cases that are vague and represent multi-factorial diagnostic dilemmas such as hypotension and hypoxemia. The ultimate goal is to strengthen patient safety by providing guidance for improving EM content, use, and training protocols.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (anesthesiologists, surgeons, nurses) participating in the crisis management curriculum at each participating simulation site

Exclusion Criteria:

* Those unwilling to be recorded during the simulation scenario

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Correct Diagnosis identified during the simulation by the participants through a grading scale tool | through scenario completion, an average of 1 hour

SECONDARY OUTCOMES:
Clinical actions taken during the scenario evaluated by a grading scale tool | through scenario completion, an average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Richard Urman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts